CLINICAL TRIAL: NCT00082745
Title: Key Adverse Events After Childhood Cancer
Brief Title: Genetic Analysis in Identifying Late-Occurring Complications in Childhood Cancer Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE03N1; COG-ALTE03N1 (CTRP (Clinical Trial Reporting Program)); CDR0000360708; ALTE03N1 (Other: Childrens Oncology Group); ALTE03N1 (Other: CTEP); U10CA180886 (NIH); U10CA095861 (NIH); UG1CA189955 (NIH); UG1CA189958 (NIH); NCT00228787 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Childhood Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and saliva

GROUPS / COHORTS (1):
- Observational (genetic analysis): DNA from peripheral blood or saliva sample of patients is analyzed for the presence of polymorphisms in genes associated with an increased risk of late-occurring complications.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies cancer survivors to identify those who are at increased risk of developing late-occurring complications after undergoing treatment for childhood cancer. A patient's genes may affect the risk of developing complications, such as congestive heart failure, avascular necrosis, stroke, and second cancer, years after undergoing cancer treatment. Genetic studies may help doctors identify survivors of childhood cancer who are more likely to develop late complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify key adverse events developing in patients (cases) with a primary cancer diagnosed at age 21 or younger.

II. To characterize the key adverse events with respect to the nature of the primary malignancy (pathology, stage) and coded details of the therapeutic protocol.

III. To identify treatment-related and demographic risk factors through a direct comparison of the case-group and controls identified from the remaining patients with the same primary diagnosis.

IV. To compare the frequency of mutations or polymorphisms in specific candidate genes in cases and controls, using constitutional deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) from the cases and controls.

V. To explore the role and nature of gene-environment interaction in the development of key adverse events.

OUTLINE:

DNA and RNA from peripheral blood or saliva sample of patients is analyzed for the presence of polymorphisms in genes associated with an increased risk of late-occurring complications.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA - CASES
* Diagnosis of primary cancer at age 21 or younger, irrespective of current age
* No prior history of allogeneic (non-autologous) hematopoietic cell transplant
* Development of one of the following key adverse events at any time following initiation of cancer therapy:

  * Cardiac dysfunction; please note: case enrollment has been closed due to achievement of target accrual
  * Ischemic stroke (IS)
  * Subsequent malignant neoplasm (SMN)
  * Avascular necrosis (AVN); please note: case enrollment has been closed due to achievement of target accrual
* Submission of a blood specimen (or in certain cases a saliva specimen) to the Coordinating Center at the University of Alabama at Birmingham as per the requirements; please note: if a patient is currently receiving active cancer treatment, it is preferable to obtain the blood sample at a time when the patient's white blood cell (WBC) is > 2,000
* Written informed consent from the patient and/or the patient's legally authorized guardian
* In active follow up by a COG institution; active follow up will be defined as date of last visit or contact by a COG institution within the past 24 months; any type of contact, including contact specifically for participation in ALTE03N1, qualifies as active follow-up; please note: treatment on a COG (or legacy group) therapeutic protocol for the primary cancer is NOT required
* ELIGIBILITY CRITERIA - CONTROLS
* CONTROL: Diagnosis of primary cancer at age 21 or younger, irrespective of current age
* CONTROLS: No prior history of allogeneic (non-autologous) hematopoietic cell transplant
* CONTROLS: No clinical evidence of any of the following key adverse events:

  * Cardiac dysfunction (CD); please note: if a patient is currently receiving active cancer treatment, it is preferable to obtain the blood sample at a time when the patient's WBC is > 2,000
  * Ischemic stroke (IS)
  * Avascular necrosis (AVN)
  * Subsequent malignant neoplasm (SMN)
* CONTROLS: Submission of a blood specimen (or in certain cases a saliva specimen) to the Coordinating Center Laboratory at the University of Alabama at Birmingham as per the requirements
* CONTROLS: Written informed consent from the patient and/or the patient's legally authorized guardian
* CONTROLS: In active follow up by a COG institution; active follow up will be defined as date of last visit or contact by a COG institution within the past 24 months; any type of contact, including contact specifically for participation in ALTE03N1, qualifies as active follow-up; please note: treatment on a COG (or legacy group) therapeutic protocol for the primary cancer is NOT required

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in active follow-up with key adverse events identified by Children's Oncology Group (COG) institutions
Sampling Method: Non-Probability Sample
Enrollment: 3885 (Estimated)
Dates: Start 2004-03-25 (Actual); Primary Completion 2004-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events (cardiac dysfunction, AVN, ischemic stroke, and SMN using a matched case-control) | Up to 1 year
  Epidemiological, clinical and laboratory variables will be tested for their association with key adverse events. McNemar's test for paired data will be used to compare the unmatched general characteristics of cases and controls.
Frequency of mutations or polymorphisms in specific candidate genes in cases and controls | Up to 1 year
  Allele frequencies will be estimated by the gene counting method, and the chi-square test will be used to check for departures from Hardy-Weinberg equilibrium.
Crude disease-exposure | Up to 1 year
  The crude disease-exposure association will be determined by estimating the OR and its 95% confidence interval (CI). This will be done by univariate conditional logistic regression, to account for the matched design. The significance of the OR will be assessed by the Wald test. Backward stepwise regression procedures will be used to develop the final multivariate model and possible interactions will be examined. The fit of the model will be assessed by the logistic regression diagnostics procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, Principal Investigator — Children's Oncology Group
Locations (156):
- United States (134):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee State University, Johnson City, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Swiss Pediatric Oncology Group - Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Singh P, Zhou L, Shah DA, Cejas RB, Crossman DK, Jouni M, Magdy T, Wang X, Sharafeldin N, Hageman L, McKenna DE, Horvath S, Armenian SH, Balis FM, Hawkins DS, Keller FG, Hudson MM, Neglia JP, Ritchey AK, Ginsberg JP, Landier W, Burridge PW, Bhatia S. Identification of novel hypermethylated or hypomethylated CpG sites and genes associated with anthracycline-induced cardiomyopathy. Sci Rep. 2023 Aug 4;13(1):12683. doi: 10.1038/s41598-023-39357-2. PMID 37542143
- [Derived] Wang X, Sun CL, Quinones-Lombrana A, Singh P, Landier W, Hageman L, Mather M, Rotter JI, Taylor KD, Chen YD, Armenian SH, Winick N, Ginsberg JP, Neglia JP, Oeffinger KC, Castellino SM, Dreyer ZE, Hudson MM, Robison LL, Blanco JG, Bhatia S. CELF4 Variant and Anthracycline-Related Cardiomyopathy: A Children's Oncology Group Genome-Wide Association Study. J Clin Oncol. 2016 Mar 10;34(8):863-70. doi: 10.1200/JCO.2015.63.4550. Epub 2016 Jan 25. PMID 26811534